CLINICAL TRIAL: NCT03106129
Title: Opioid Requirements Post Discharge of Patients Having Total Knee Arthroplasty (TKA)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 309-2016
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Knee Arthropathy; Opioid Use; Pain; Rehabilitation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total knee arthroplasty (TKA) may result in significant postoperative pain. The majority of these patients are prescribed opioids for the management of postoperative pain. Recent evidence has highlighted that postoperative opioids are being over-prescribed resulting in opioid misuse and abuse. Over-prescribing also results in a significant financial cost. This prospective observational study was designed to determine the mean amount of opioid required after TKA. This data can be used in the future as a guide to change our current practice of prescribing with the aim to reduce over-prescription.

DETAILED DESCRIPTION:
Over prescription of opioids is currently a National epidemic . There is a call for action to address this problem urgently and anesthesiologists are well positioned to participate and lead through research to educate medical practitioners of how to prescribe the optimal dose with the ultimate goal of improved patient's safety.

Total knee arthroplasy (TKA) and total hip arthroplasty (THA) may result in significant and sustained postoperative pain. For optimal pain control, faster recovery, and better functional rehabilitation, these patients are prescribed opioids in addition to analgesic adjuncts in hospital and after discharge from the hospital. This practice stems from much evidence that demonstrated a propensity for moderate and severe pain of 52% and 16% respectively up to 30 days post discharge in patients undergoing THA and TKA.

These patients are prescribed opioids upon discharge from the hospital to control pain and to enhance optimal rehabilitation. The discharge prescription is often based on a surgeon's judgment and past experience. Furthermore, more than 50% of patients may receive suboptimal pain control resulting in pain in the early postoperative period. On the other hand, recent studies have shown that opioids are often over-prescribed. This practice not only results in a significant financial cost, but also represents a potential reservoir for opioid misuse and abuse. In Canada, the rate of dispensing high-dose opioid formulations (greater than 200mg morphine equivalents per day) increased 23.0%, from 781 units per 1000 population in 2006 to 961 units per 1000 population in 2011. Excessive opioid prescriptions can lead to excessive morbidity and mortality as evidenced in the United States where 16 917 (74%) of the 22,810 deaths relating to pharmaceutical overdose involved opioid analgesics. With respect to the financial burden, in the United States in 2007, prescription opioid abuse costs were $55.7 billion of which 45% were healthcare costs (e.g., abuse treatment).

To the author's knowledge there are no widely used objective tools or guidelines to instruct patients in self-administering opioids post-discharge or to help surgeons to avoid over or under prescribing. This may contribute to either over-dosing with opioid related side effects, or under-dosing with inadequate analgesia and rehabilitation.

In this prospective observational study we plan to determine the mean amount of opioid required post discharge after TKA that correlates with good pain management and rehabilitation outcomes. The mean amount of opioid consumed could be used in the future to guide physicians to practice proper opioid prescribing post discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Having an elective total knee replacement done at Sunnybrook Holland Orthopaedic and Arthritic Centre.
* All participants must speak English and have no communication barriers.

Exclusion Criteria:

* If you are taking >10mg morphine equivalents per day
* Deemed incompetent to be able to self prescribe opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants must be 18 years or older and are undergoing an elective total knee arthroplasty at Sunnybrook Holland Orthopaedic and Arthritic Centre. All participants must speak English and be able to receive phone calls once a week for 6 weeks after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-02-09 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The amount of opioid analgesics used and the number remaining | 6 weeks after surgery
  A member of the research team will contact the participant weekly after their surgery. Over the phone the team member will collect the total amount of opioid taken and the total amount of opioid remaining.

SECONDARY OUTCOMES:
The amount of non-opioid analgesics consumed | 6 weeks after surgery
  The team member will contact the participant weekly to ask about the number of other non-opioid analgesics consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Imad Awad, MBChB, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buckley N. The prescription opioid epidemic: a call to action for our profession. Can J Anaesth. 2016 Jan;63(1):8-11. doi: 10.1007/s12630-015-0521-x. Epub 2015 Oct 23. No abstract available. PMID 26497722
- [Background] Alam A, Juurlink DN. The prescription opioid epidemic: an overview for anesthesiologists. Can J Anaesth. 2016 Jan;63(1):61-8. doi: 10.1007/s12630-015-0520-y. Epub 2015 Oct 27. PMID 26507535
- [Background] Kharasch ED, Brunt LM. Perioperative Opioids and Public Health. Anesthesiology. 2016 Apr;124(4):960-5. doi: 10.1097/ALN.0000000000001012. No abstract available. PMID 26808634
- [Background] Barrington JW, Halaszynski TM, Sinatra RS, Expert Working Group On Anesthesia And Orthopaedics Critical Issues In Hip And Knee Replacement Arthroplasty FT. Perioperative pain management in hip and knee replacement surgery. Am J Orthop (Belle Mead NJ). 2014 Apr;43(4 Suppl):S1-S16. PMID 24911869
- [Background] Roberts M, Brodribb W, Mitchell G. Reducing the pain: a systematic review of postdischarge analgesia following elective orthopedic surgery. Pain Med. 2012 May;13(5):711-27. doi: 10.1111/j.1526-4637.2012.01359.x. Epub 2012 Apr 11. PMID 22494470
- [Background] Andersen LO, Gaarn-Larsen L, Kristensen BB, Husted H, Otte KS, Kehlet H. Subacute pain and function after fast-track hip and knee arthroplasty. Anaesthesia. 2009 May;64(5):508-13. doi: 10.1111/j.1365-2044.2008.05831.x. PMID 19413820
- [Background] Rawal N. Postoperative pain treatment for ambulatory surgery. Best Pract Res Clin Anaesthesiol. 2007 Mar;21(1):129-48. doi: 10.1016/j.bpa.2006.11.005. PMID 17489224
- [Background] Maheshwari AV, Blum YC, Shekhar L, Ranawat AS, Ranawat CS. Multimodal pain management after total hip and knee arthroplasty at the Ranawat Orthopaedic Center. Clin Orthop Relat Res. 2009 Jun;467(6):1418-23. doi: 10.1007/s11999-009-0728-7. Epub 2009 Feb 13. PMID 19214642
- [Background] Rodgers J, Cunningham K, Fitzgerald K, Finnerty E. Opioid consumption following outpatient upper extremity surgery. J Hand Surg Am. 2012 Apr;37(4):645-50. doi: 10.1016/j.jhsa.2012.01.035. Epub 2012 Mar 10. PMID 22410178
- [Background] Manchikanti L, Fellows B, Ailinani H, Pampati V. Therapeutic use, abuse, and nonmedical use of opioids: a ten-year perspective. Pain Physician. 2010 Sep-Oct;13(5):401-35. PMID 20859312
- [Background] Gomes T, Mamdani MM, Paterson JM, Dhalla IA, Juurlink DN. Trends in high-dose opioid prescribing in Canada. Can Fam Physician. 2014 Sep;60(9):826-32. PMID 25217680
- [Background] Birnbaum HG, White AG, Schiller M, Waldman T, Cleveland JM, Roland CL. Societal costs of prescription opioid abuse, dependence, and misuse in the United States. Pain Med. 2011 Apr;12(4):657-67. doi: 10.1111/j.1526-4637.2011.01075.x. Epub 2011 Mar 10. PMID 21392250
- [Background] Skinner HB, Shintani EY. Results of a multimodal analgesic trial involving patients with total hip or total knee arthroplasty. Am J Orthop (Belle Mead NJ). 2004 Feb;33(2):85-92; discussion 92. PMID 15005598
- [Background] Wainwright AV, Kennedy DM, Stratford PW. The Group Experience: Remodelling Outpatient Physiotherapy after Knee Replacement Surgery. Physiother Can. 2015 Fall;67(4):350-6. doi: 10.3138/ptc.2014-44. PMID 27504034
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543